CLINICAL TRIAL: NCT03130634
Title: The Efficacy of Silymarin as Adjuvant Therapy on Colorectal Cancer Patients Undergoing FOLFIRI Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jaw-Yuan Wang, MD, PhD, Professor, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KMUHIRB-F(II)-20160038
Record Dates: First submitted 2017-04-22; First posted 2017-04-26 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Metastatic Colorectal Cancer
Keywords: CPT-11(irinotecan); silymarin; GI toxicity
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Silymarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prescription of silymarin (Experimental): During six cycles of FOLFIRI chemotherapy, the patients will take silymarin (150mg) three times daily from day 1 to day 7 during one cycle of treatment.
  Interventions: Drug: Silymarin
- control (No Intervention): During six cycles of FOLFIRI chemotherapy, the patients will not take silymarin during chemotherapy

INTERVENTIONS:
Drug: Silymarin — During six cycles of FOLFIRI chemotherapy, the patients will take silymarin (150mg) three times daily from day 1 to day 7 during one cycle of treatment.
  Arms: prescription of silymarin

SUMMARY:
Primary objectives: Use both listed and relatively safe drug, Silymarin,s to improve the intestinal side effect of the patients undergoing FOLFIRI chemotherapy.

DETAILED DESCRIPTION:
Primary Objective:

Use both listed and relatively safe drug, Silymarin, to improve the intestinal side effect of the patients undergoing FOLFIRI chemotherapy.

Patient Selection and Enrollment:

Number of Subjects: Eligible patients will be randomized in 2 arms in the ratio of 1:1, to reach approximately 70 patients in total.

Plan of the Study:

Study Design This is an open-label, randomized, comparative, double arm, single center study to assess efficacy of Silymarin as adjuvant therapy on metastatic colorectal cancer patients undergoing FOLFIRI chemotherapy in Taiwan.

Subject Number Eligible patients will be randomized in 2 arms in the ratio of 1:1, to reach approximately 70 patients in total.

Study Schedule Study date: the time getting approval letter issued by both regulatory authority and institutional review board (IRB) Duration of study: From the date of the IRB was approved till the 70th patient was collected.

Duration of Enrollment: From the date of the IRB was approved till the 70th patient was collected.

Duration of treatment: From the 1st patient starting chemotherapy till the 70th patient finishing the 6th cycle chemotherapy.

Duration of follow-up: From the 1st patient starting chemotherapy till 3 months after the 70th patient finishing the 6th cycle chemotherapy

ELIGIBILITY:
Inclusion Criteria:

1. The patient who is between 20 to 80 years old
2. The patient who is diagnosed metastatic colorectal cancer and received chemotherapy with FOLFIRI regimen
3. The female patient should not be pregnant or breast-feeding
4. The patient who has no severe co-morbidity, such as cardiovascular, cerebrovascular, malignant hypertension, renal and hepatobiliary disease.
5. The patient who has no associated drug allergy to this trial.
6. The patient who is in compliance with prescribed medication.
7. The patient who is willing to sign the permit of the clinical trial.

Exclusion Criteria:

1. The patients who do not meet the main inclusion criteria or are not willing to sign the permit.
2. The patient who has viral hepatitis or carrier with impaired liver function.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
GI associated adverse events | 3 months
  Response rate and grades of GI associated adverse events (AEs) according to the Response Evaluation Criteria in Solid Tumors (version 1.1)

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-Ho Memorial Hospital, Kaohsiung Medical University:, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided